CLINICAL TRIAL: NCT03220165
Title: An Open-Label, Single-Radiolabeled Dose, Non-Randomized Study to Determine the Mass Balance of [14C] MGL-3196
Brief Title: Radiolabeled Study to Determine the Mass Balance of [14C] MGL-3196
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGL-3196-07
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — resmetirom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): MGL-3196
  Interventions: Drug: MGL-3196

INTERVENTIONS:
Drug: MGL-3196 — oral, 100 mg
  Other Names: VIA-3196

SUMMARY:
The purpose of this study is determine in healthy males how MGL-3196 is metabolized using a radio-labeled version of MGL-3196.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily consents to participate and provides written informed consent.
* Is a male.
* Is between 18 and 55 years of age (inclusive).
* Has a body mass index (BMI) between 18 and 32 kg/m2 (inclusive), and weighs a minimum of 50 kg.
* Is willing and able to remain in the study unit for the entire duration of the confinement periods
* Is willing to eat entire meals and snacks provided during confinement at the research facility; and understand that the diet will include foods with high fiber content and possibly prune juice.
* Is willing to have collected all urine and fecal samples for the duration of the study period as required.
* Is willing to use a waterless commode located in a designated dry room for urine and feces collection for the duration of the study period as required.
* Is willing to abstain from showering for the first 72 hours after administration of [14C] MGL-3196. After the restriction from showering is lifted, must be willing to provide a urine sample prior to showering for the remainder of the confinement period.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* A clinically significant abnormal finding on the physical exam, medical history, electrocardiogram (ECG), or clinical laboratory results at screening.
* Thyroid stimulating hormone test at screening outside the normal range. Repeat testing is allowed once at the discretion of the Investigator.
* Current or recent (<6 months) hepatobiliary disease; or AST, ALT or direct bilirubin greater than the upper limit of reference range at screening. Repeat testing is allowed once at the discretion of the Investigator.
* Elevated CK at screening (one repeat test allowed).
* History of Gilbert's syndrome.
* Pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study drug.
* Abnormal screening ECG: including machine-read QTcF >450 msec (confirmed by manual over read), QRS >110 msec, intermittent bundle branch block, frequent premature atrial or premature ventricular contractions, or any rhythm other than normal sinus rhythm which is interpreted by the Investigator to be clinically significant.
* History of sensitivity to a similar study drug (e.g., Karo Bio KB2115 or Metabasis MB7811), or a history of important drug or other allergy (except for untreated, asymptomatic seasonal allergies at time of dosing) unless deemed not clinically significant by the Investigator.
* History of sensitivity to thyroid medication.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has participated in a standard radiolabeled clinical trial within the last 12 months prior to the first dose of study medication or a micro tracer clinical trial within the last 3 months prior to the first dose of study medication.
* Has participated in another clinical trial (randomized subjects only) within 30 days prior to the first dose of study medication.
* Use of any over-the-counter (OTC) medication (including nutritional or dietary supplements, herbal preparations, vitamins, or acetaminophen) within 7 days prior to the first dose of study medication until the end of study visit without evaluation and approval by the Investigator.
* Use of any prescription medication from 14 days prior to the first dose of study medication until the end-of-study visit without evaluation and approval by the Investigator.
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days prior to the first dose of study medication, and that, in the Investigator's judgment, may impact subject safety or the validity of the study results.
* Blood or plasma donation within 30 days prior to the first dose of study medication until the end-of-study visit. It is recommended that blood/plasma donations not be made for at least 30 days after the end-of-study visit.
* Smoking or use of tobacco- or nicotine-containing products within 60 days prior to the first dose of study medication until the end-of-study visit.
* Consumption of beverages or foods that contain grapefruit, poppy seeds, broccoli, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to the first dose of study medication until the end-of-study visit. Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study Investigator based on the potential for interaction with the study drug.
* Has any prior history of substance abuse or treatment (including alcohol).
* History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months prior to screening.
* Use of alcohol within 24 hours prior to dosing and throughout the study.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates) or cotinine.
* Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
* Excessive caffeine intake (>3 cups of coffee/day or equivalent).
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical disease (e.g., infectious disease) must not be enrolled.
* Any other sound medical, psychiatric, and /or social reason as determined by the Investigator.
* Has irregular bowel habits. ("Irregular" being defined for the purpose of this study as NOT having a bowel movement at least every 2 days.)
* Has been exposed to radiation, including dental or medical imaging such as X-ray or tomography, in the 6 months prior to dose administration.
* Has been involved in an occupation that requires monitoring for radiation exposure (eg, X-ray technician).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-06 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-03 (Actual)

PRIMARY OUTCOMES:
Mass Balance of [14C] MGL-3196 | Approximately 10 Days
  Measurement of the total radioactivity collected from blood, urine, and feces

CONTACTS AND LOCATIONS:
Overall Officials: George Ate, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No